CLINICAL TRIAL: NCT02270242
Title: Ticagrelor With Aspirin or Alone in High-Risk Patients After Coronary Intervention
Acronym: TWILIGHT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Roxana Mehran, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GCO 14-1383
Record Dates: First submitted 2014-10-15; First posted 2014-10-21 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Cardiovascular Disease; Interventional Cardiology
Keywords: PCI; DAPT; ticagrelor; aspirin
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Aspirin; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aspirin + Ticagrelor (Active Comparator): enteric coated aspirin 81mg-100mg daily p.o. for 12 months and ticagrelor 90mg tablet bid for 12 months
  Interventions: Drug: Aspirin; Drug: ticagrelor
- Placebo + Ticagrelor (Placebo Comparator): placebo pill daily p.o. for 12 months - match for enteric coated aspirin 81mg-100mg and ticagrelor 90mg tablet bid for 12 months
  Interventions: Drug: Placebo; Drug: ticagrelor

INTERVENTIONS:
Drug: Aspirin
  Other Names: Ecotrin
  Arms: Aspirin + Ticagrelor
Drug: Placebo
  Arms: Placebo + Ticagrelor
Drug: ticagrelor
  Other Names: Brilinta; Brilique

SUMMARY:
The purpose of this study is to compare the use of ticagrelor alone versus ticagrelor and aspirin together. Both ticagrelor and aspirin stop platelets from sticking together and forming a blood clot that could block blood flow to the heart. This study will look to determine the effectiveness and safety of ticagrelor alone, compared to ticagrelor plus aspirin in reducing clinically relevant bleeding and in reducing ischemic adverse events among high-risk patients who have had a percutaneous intervention with at least one drug-eluting stent. A patient is considered high-risk if they meet certain clinical and/or anatomic criteria.

Up to 9000 subjects will be enrolled at the time of their index PCI. Subjects meeting randomization eligibility criteria at 3 months post enrollment will be randomized to either ticagrelor plus aspirin or ticagrelor plus placebo for an additional 12 months. Follow-up clinic visits will be performed at 3 months, 9 months and 15 months post enrollment.

DETAILED DESCRIPTION:
This is a multicenter, prospective, blinded dual-arm study. Up to 9000 high-risk patients who have undergone successful PCI with at least one locally approved drug eluting stent discharged on DAPT with aspirin and ticagrelor of at least 3 months intended duration from centers still to be determined in the U.S., Canada, Europe and Asia. The primary objective of this study is to determine the impact of antiplatelet monotherapy with ticagrelor alone versus DAPT with ticagrelor plus aspirin for 12 months in reducing clinically relevant bleeding (efficacy) among high-risk patients undergoing PCI who have completed a 3-month course of aspirin plus ticagrelor. The secondary objective of this study is to determine the impact of antiplatelet monotherapy with ticagrelor alone versus DAPT with ticagrelor plus aspirin for 12 months in reducing major ischemic adverse events (safety) among high-risk patients undergoing PCI who have completed a 3-month course of aspirin plus ticagrelor.

Exploratory objectives include assessing the comparative safety and efficacy of the different DAPT regimens for individual components of the primary efficacy and secondary safety objectives.

The primary analysis for TWILIGHT will be performed independently by the London School of Hygiene and Tropical Medicine

ELIGIBILITY:
Inclusion Criteria:

* High-risk patients who have undergone successful PCI with at least one locally approved drug eluting stent discharged on DAPT with aspirin and ticagrelor of at least 3 months intended duration will be eligible for the TWILIGHT study.
* Enrollment into the study will require meeting at least one clinical inclusion, one angiographic inclusion and none of the exclusion criteria.

Clinical Inclusion Criteria:

* Adult patients ≥ 65 years of age
* Female gender
* Troponin Positive acute coronary syndrome
* Established vascular disease defined as previous MI, documented PAD or CAD/PAD revascularization
* Diabetes mellitus treated with medications (oral hypoglycemic, subcutaneous injection of insulin)
* Chronic kidney disease defined as an estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73m2 or creatinine clearance (CrCl) < 60 ml/min

Angiographic Inclusion Criteria:

* Multivessel coronary artery disease
* Target lesion requiring total stent length >30 mm
* Thrombotic target lesion(s)
* Bifurcation lesions with Medina X,1,1 classification requiring at least 2 stents
* Left main (≥50%) or proximal LAD (≥70%) lesion
* Calcified target lesion(s) requiring atherectomy

Exclusion Criteria:

* Under 18 years of age
* Contraindication to aspirin
* Contraindication to ticagrelor
* Planned surgery within 90 days
* Planned coronary revascularization (surgical or percutaneous) within 90 days
* Need for chronic oral anticoagulation
* Prior stroke
* Dialysis-dependent renal failure
* Active bleeding or extreme-risk for major bleeding (e.g. active peptic ulcer disease, gastrointestinal pathology with a raised risk for bleeding, malignancies with a raised risk for bleeding)
* Salvage PCI or STEMI presentation.
* Liver cirrhosis
* Life expectancy < 1 year
* Unable or unwilling to provide informed consent
* Women of child bearing potential. Defined: a woman is considered potential (WOBCP) following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. a postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Fibrinolytic therapy within 24 hours of index PCI
* Concomitant therapy with a strong cytochrome P-450 3A inhibitor or inducer
* Platelet count < 100,000 mm3
* Requiring ongoing treatment with aspirin ≥ 325 mg daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9006 (Actual)
Dates: Start 2015-07; Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Mehran, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Usman Baber, MD, Study Director — Icahn School of Medicine at Mount Sinai; Roxana Mehran, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS, Smith SC Jr, Jacobs AK, Halperin JL, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non ST-Elevation Myocardial Infarction); American College of Emergency Physicians; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; American Association of Cardiovascular and Pulmonary Rehabilitation; Society for Academic Emergency Medicine. ACC/AHA 2007 guidelines for the management of patients with unstable angina/non ST-elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non ST-Elevation Myocardial Infarction): developed in collaboration with the American College of Emergency Physicians, the Society for Cardiovascular Angiography and Interventions, and the Society of Thoracic Surgeons: endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation and the Society for Academic Emergency Medicine. Circulation. 2007 Aug 14;116(7):e148-304. doi: 10.1161/CIRCULATIONAHA.107.181940. Epub 2007 Aug 6. No abstract available. PMID 17679616
- [Background] Antman EM, Anbe DT, Armstrong PW, Bates ER, Green LA, Hand M, Hochman JS, Krumholz HM, Kushner FG, Lamas GA, Mullany CJ, Ornato JP, Pearle DL, Sloan MA, Smith SC Jr, Alpert JS, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Gregoratos G, Halperin JL, Hiratzka LF, Hunt SA, Jacobs AK; American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 1999 Guidelines for the Management of Patients With Acute Myocardial Infarction). ACC/AHA guidelines for the management of patients with ST-elevation myocardial infarction--executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 1999 Guidelines for the Management of Patients With Acute Myocardial Infarction). Circulation. 2004 Aug 3;110(5):588-636. doi: 10.1161/01.CIR.0000134791.68010.FA. No abstract available. PMID 15289388
- [Background] King SB 3rd, Smith SC Jr, Hirshfeld JW Jr, Jacobs AK, Morrison DA, Williams DO, Feldman TE, Kern MJ, O'Neill WW, Schaff HV, Whitlow PL; ACC/AHA/SCAI; Adams CD, Anderson JL, Buller CE, Creager MA, Ettinger SM, Halperin JL, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura R, Page RL, Riegel B, Tarkington LG, Yancy CW. 2007 focused update of the ACC/AHA/SCAI 2005 guideline update for percutaneous coronary intervention: a report of the American College of Cardiology/American Heart Association Task Force on Practice guidelines. J Am Coll Cardiol. 2008 Jan 15;51(2):172-209. doi: 10.1016/j.jacc.2007.10.002. No abstract available. PMID 18191745
- [Background] Dupont AG, Gabriel DA, Cohen MG. Antiplatelet therapies and the role of antiplatelet resistance in acute coronary syndrome. Thromb Res. 2009 May;124(1):6-13. doi: 10.1016/j.thromres.2009.01.014. Epub 2009 Mar 25. PMID 19324398
- [Background] Geisler T, Zurn C, Simonenko R, Rapin M, Kraibooj H, Kilias A, Bigalke B, Stellos K, Schwab M, May AE, Herdeg C, Gawaz M. Early but not late stent thrombosis is influenced by residual platelet aggregation in patients undergoing coronary interventions. Eur Heart J. 2010 Jan;31(1):59-66. doi: 10.1093/eurheartj/ehp402. Epub 2009 Oct 6. PMID 19812059
- [Background] Hochholzer W, Trenk D, Bestehorn HP, Fischer B, Valina CM, Ferenc M, Gick M, Caputo A, Buttner HJ, Neumann FJ. Impact of the degree of peri-interventional platelet inhibition after loading with clopidogrel on early clinical outcome of elective coronary stent placement. J Am Coll Cardiol. 2006 Nov 7;48(9):1742-50. doi: 10.1016/j.jacc.2006.06.065. Epub 2006 Oct 17. PMID 17084243
- [Background] Marcucci R, Gori AM, Paniccia R, Giusti B, Valente S, Giglioli C, Buonamici P, Antoniucci D, Abbate R, Gensini GF. Cardiovascular death and nonfatal myocardial infarction in acute coronary syndrome patients receiving coronary stenting are predicted by residual platelet reactivity to ADP detected by a point-of-care assay: a 12-month follow-up. Circulation. 2009 Jan 20;119(2):237-42. doi: 10.1161/CIRCULATIONAHA.108.812636. Epub 2008 Dec 31. PMID 19118249
- [Background] Jernberg T, Payne CD, Winters KJ, Darstein C, Brandt JT, Jakubowski JA, Naganuma H, Siegbahn A, Wallentin L. Prasugrel achieves greater inhibition of platelet aggregation and a lower rate of non-responders compared with clopidogrel in aspirin-treated patients with stable coronary artery disease. Eur Heart J. 2006 May;27(10):1166-73. doi: 10.1093/eurheartj/ehi877. Epub 2006 Apr 18. PMID 16621870
- [Background] Wallentin L, Varenhorst C, James S, Erlinge D, Braun OO, Jakubowski JA, Sugidachi A, Winters KJ, Siegbahn A. Prasugrel achieves greater and faster P2Y12receptor-mediated platelet inhibition than clopidogrel due to more efficient generation of its active metabolite in aspirin-treated patients with coronary artery disease. Eur Heart J. 2008 Jan;29(1):21-30. doi: 10.1093/eurheartj/ehm545. Epub 2007 Nov 30. PMID 18055486
- [Background] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Background] van Giezen JJ, Humphries RG. Preclinical and clinical studies with selective reversible direct P2Y12 antagonists. Semin Thromb Hemost. 2005 Apr;31(2):195-204. doi: 10.1055/s-2005-869525. PMID 15852223
- [Background] Husted S, Emanuelsson H, Heptinstall S, Sandset PM, Wickens M, Peters G. Pharmacodynamics, pharmacokinetics, and safety of the oral reversible P2Y12 antagonist AZD6140 with aspirin in patients with atherosclerosis: a double-blind comparison to clopidogrel with aspirin. Eur Heart J. 2006 May;27(9):1038-47. doi: 10.1093/eurheartj/ehi754. Epub 2006 Feb 13. PMID 16476694
- [Background] Storey RF, Husted S, Harrington RA, Heptinstall S, Wilcox RG, Peters G, Wickens M, Emanuelsson H, Gurbel P, Grande P, Cannon CP. Inhibition of platelet aggregation by AZD6140, a reversible oral P2Y12 receptor antagonist, compared with clopidogrel in patients with acute coronary syndromes. J Am Coll Cardiol. 2007 Nov 6;50(19):1852-6. doi: 10.1016/j.jacc.2007.07.058. Epub 2007 Oct 23. PMID 17980251
- [Background] Alexopoulos D, Galati A, Xanthopoulou I, Mavronasiou E, Kassimis G, Theodoropoulos KC, Makris G, Damelou A, Tsigkas G, Hahalis G, Davlouros P. Ticagrelor versus prasugrel in acute coronary syndrome patients with high on-clopidogrel platelet reactivity following percutaneous coronary intervention: a pharmacodynamic study. J Am Coll Cardiol. 2012 Jul 17;60(3):193-9. doi: 10.1016/j.jacc.2012.03.050. PMID 22789884
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Baber U, Mehran R, Sharma SK, Brar S, Yu J, Suh JW, Kim HS, Park SJ, Kastrati A, de Waha A, Krishnan P, Moreno P, Sweeny J, Kim MC, Suleman J, Pyo R, Wiley J, Kovacic J, Kini AS, Dangas GD. Impact of the everolimus-eluting stent on stent thrombosis: a meta-analysis of 13 randomized trials. J Am Coll Cardiol. 2011 Oct 4;58(15):1569-77. doi: 10.1016/j.jacc.2011.06.049. Epub 2011 Sep 14. PMID 21924575
- [Background] Feres F, Costa RA, Abizaid A, Leon MB, Marin-Neto JA, Botelho RV, King SB 3rd, Negoita M, Liu M, de Paula JE, Mangione JA, Meireles GX, Castello HJ Jr, Nicolela EL Jr, Perin MA, Devito FS, Labrunie A, Salvadori D Jr, Gusmao M, Staico R, Costa JR Jr, de Castro JP, Abizaid AS, Bhatt DL; OPTIMIZE Trial Investigators. Three vs twelve months of dual antiplatelet therapy after zotarolimus-eluting stents: the OPTIMIZE randomized trial. JAMA. 2013 Dec 18;310(23):2510-22. doi: 10.1001/jama.2013.282183. PMID 24177257
- [Background] Valgimigli M, Campo G, Monti M, Vranckx P, Percoco G, Tumscitz C, Castriota F, Colombo F, Tebaldi M, Fuca G, Kubbajeh M, Cangiano E, Minarelli M, Scalone A, Cavazza C, Frangione A, Borghesi M, Marchesini J, Parrinello G, Ferrari R; Prolonging Dual Antiplatelet Treatment After Grading Stent-Induced Intimal Hyperplasia Study (PRODIGY) Investigators. Short- versus long-term duration of dual-antiplatelet therapy after coronary stenting: a randomized multicenter trial. Circulation. 2012 Apr 24;125(16):2015-26. doi: 10.1161/CIRCULATIONAHA.111.071589. Epub 2012 Mar 21. PMID 22438530
- [Background] Brar SS, Kim J, Brar SK, Zadegan R, Ree M, Liu IL, Mansukhani P, Aharonian V, Hyett R, Shen AY. Long-term outcomes by clopidogrel duration and stent type in a diabetic population with de novo coronary artery lesions. J Am Coll Cardiol. 2008 Jun 10;51(23):2220-7. doi: 10.1016/j.jacc.2008.01.063. PMID 18534267
- [Background] Gwon HC, Hahn JY, Park KW, Song YB, Chae IH, Lim DS, Han KR, Choi JH, Choi SH, Kang HJ, Koo BK, Ahn T, Yoon JH, Jeong MH, Hong TJ, Chung WY, Choi YJ, Hur SH, Kwon HM, Jeon DW, Kim BO, Park SH, Lee NH, Jeon HK, Jang Y, Kim HS. Six-month versus 12-month dual antiplatelet therapy after implantation of drug-eluting stents: the Efficacy of Xience/Promus Versus Cypher to Reduce Late Loss After Stenting (EXCELLENT) randomized, multicenter study. Circulation. 2012 Jan 24;125(3):505-13. doi: 10.1161/CIRCULATIONAHA.111.059022. Epub 2011 Dec 16. PMID 22179532
- [Background] Chirumamilla AP, Maehara A, Mintz GS, Mehran R, Kanwal S, Weisz G, Hassanin A, Hakim D, Guo N, Baber U, Pyo R, Moses JW, Fahy M, Kovacic JC, Dangas GD. High platelet reactivity on clopidogrel therapy correlates with increased coronary atherosclerosis and calcification: a volumetric intravascular ultrasound study. JACC Cardiovasc Imaging. 2012 May;5(5):540-9. doi: 10.1016/j.jcmg.2011.12.019. PMID 22595163
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Wiviott SD, Antman EM, Gibson CM, Montalescot G, Riesmeyer J, Weerakkody G, Winters KJ, Warmke JW, McCabe CH, Braunwald E; TRITON-TIMI 38 Investigators. Evaluation of prasugrel compared with clopidogrel in patients with acute coronary syndromes: design and rationale for the TRial to assess Improvement in Therapeutic Outcomes by optimizing platelet InhibitioN with prasugrel Thrombolysis In Myocardial Infarction 38 (TRITON-TIMI 38). Am Heart J. 2006 Oct;152(4):627-35. doi: 10.1016/j.ahj.2006.04.012. PMID 16996826
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432
- [Derived] Steg PG, Nicolas J, Baber U, Sartori S, Zhang Z, Feng Y, Angiolillo DJ, Briguori C, Cohen DJ, Collier T, Dangas G, Dudek D, Escaned J, Gibson CM, Han YL, Huber K, Kastrati A, Kaul U, Marx SO, Kornowski R, Kunadian V, Vogel B, Oliva A, Mehta SR, Moliterno D, Sardella G, Krucoff M, Shlofmitz RA, Sharma S, Pocock S, Mehran R. Characterizing high-risk enrollment criteria and impact on clinical outcomes in a large randomized clinical trial: Insights from the TWILIGHT trial. Am Heart J. 2025 Aug;286:97-107. doi: 10.1016/j.ahj.2025.01.016. Epub 2025 Jan 30. PMID 39889917
- [Derived] Krucoff M, Spirito A, Baber U, Sartori S, Angiolillo DJ, Briguori C, Cohen DJ, Collier T, Dangas G, Dudek D, Escaned J, Gibson CM, Han YL, Huber K, Kastrati A, Kaul U, Kornowski R, Kunadian V, Vogel B, Mehta SR, Moliterno D, Sardella G, Shlofmitz RA, Sharma S, Steg PG, Pocock S, Mehran R. Ticagrelor with or without aspirin following percutaneous coronary intervention in high-risk patients with concomitant peripheral artery disease: A subgroup analysis of the TWILIGHT randomized clinical trial. Am Heart J. 2024 Jun;272:11-22. doi: 10.1016/j.ahj.2024.03.002. Epub 2024 Mar 6. PMID 38458371
- [Derived] Baber U, Spirito A, Sartori S, Angiolillo DJ, Briguori C, Cohen DJ, Collier T, Dangas G, Dudek D, Escaned J, Gibson CM, Han YL, Huber K, Kastrati A, Kaul U, Kornowski R, Krucoff M, Kunadian V, Vogel B, Mehta SR, Moliterno D, Sardella G, Shlofmitz RA, Sharma S, Steg PG, Pocock S, Mehran R. Clinically Driven Revascularization in High-Risk Patients Treated With Ticagrelor Monotherapy After PCI: Insights from the Randomized TWILIGHT Trial. Am J Cardiol. 2023 Dec 1;208:16-24. doi: 10.1016/j.amjcard.2023.09.008. Epub 2023 Oct 6. PMID 37806185
- [Derived] Mendieta G, Mehta S, Baber U, Angiolillo DJ, Briguori C, Cohen D, Collier T, Dangas G, Dudek D, Escaned J, Gil R, Vogel B, Cao D, Spirito A, Huber K, Kastrati A, Kaul U, Kornowski R, Krucoff MW, Kunadian V, Moliterno DJ, Ohman EM, Sardella G, Sartori S, Sharma S, Shlofmitz R, Steg PG, Han YL, Pocock S, Gibson CM, Mehran R. Bleeding and Ischemic Risks of Ticagrelor Monotherapy After Coronary Interventions. J Am Coll Cardiol. 2023 Aug 22;82(8):687-700. doi: 10.1016/j.jacc.2023.05.062. PMID 37587580
- [Derived] Spirito A, Koh WJ, Sartori S, Vogel B, Feng Y, Baber U, Nicolas J, Snyder C, Kamaleldin K, Pileggi B, Rezvanizadeh V, Sweeny J, Sharma SK, Kini A, Pocock SJ, Dangas G, Mehran R. Fatal, ischemic and bleeding risk of patients meeting the selection criteria of the TWILIGHT trial: Insights from a large PCI registry. Am Heart J. 2023 Sep;263:26-34. doi: 10.1016/j.ahj.2023.04.007. Epub 2023 Apr 23. PMID 37094668
- [Derived] Spirito A, Kastrati A, Cao D, Baber U, Sartori S, Angiolillo DJ, Briguori C, Cohen DJ, Dangas G, Dudek D, Escaned J, Gibson CM, Zhang Z, Huber K, Kaul U, Kornowski R, Kunadian V, Han YL, Mehta SR, Sardella G, Sharma S, Shlofmitz RA, Vogel B, Collier T, Pocock S, Mehran R. Ticagrelor with or without aspirin in high-risk patients with anaemia undergoing percutaneous coronary intervention: a subgroup analysis of the TWILIGHT trial. Eur Heart J Cardiovasc Pharmacother. 2023 Jun 2;9(4):328-336. doi: 10.1093/ehjcvp/pvad006. PMID 36649694
- [Derived] Han Y, Claessen BE, Chen SL, Chunguang Q, Zhou Y, Xu Y, Hailong L, Chen J, Qiang W, Zhang R, Luo S, Li Y, Zhu J, Zhao X, Cheng X, Wang J, Su X, Tao J, Sun Y, Wang G, Li Y, Bian L, Goel R, Sartori S, Zhang Z, Angiolillo DJ, Cohen DJ, Gibson CM, Kastrati A, Krucoff M, Mehta SR, Ohman EM, Steg PG, Liu Y, Dangas G, Sharma S, Baber U, Mehran R. Ticagrelor With or Without Aspirin in Chinese Patients Undergoing Percutaneous Coronary Intervention: A TWILIGHT China Substudy. Circ Cardiovasc Interv. 2022 Apr;15(4):e009495. doi: 10.1161/CIRCINTERVENTIONS.120.009495. Epub 2022 Mar 23. PMID 35317615
- [Derived] Chiarito M, Baber U, Cao D, Sharma SK, Dangas G, Angiolillo DJ, Briguori C, Cohen DJ, Dudek D, Dzavik V, Escaned J, Gil R, Hamm CW, Henry T, Huber K, Kastrati A, Kaul U, Kornowski R, Krucoff M, Kunadian V, Mehta SR, Moliterno D, Ohman EM, Oldroyd K, Sardella G, Zhongjie Z, Sartori S, Stefanini G, Shlofmitz R, Steg PG, Weisz G, Witzenbichler B, Han YL, Pocock S, Gibson CM, Mehran R. Ticagrelor Monotherapy After PCI in High-Risk Patients With Prior MI: A Prespecified TWILIGHT Substudy. JACC Cardiovasc Interv. 2022 Feb 14;15(3):282-293. doi: 10.1016/j.jcin.2021.11.005. Epub 2022 Jan 12. PMID 35033468
- [Derived] Vogel B, Baber U, Cohen DJ, Sartori S, Sharma SK, Angiolillo DJ, Farhan S, Goel R, Zhang Z, Briguori C, Collier T, Dangas G, Dudek D, Escaned J, Gil R, Han YL, Kaul U, Kornowski R, Krucoff MW, Kunadian V, Mehta SR, Moliterno D, Ohman EM, Sardella G, Witzenbichler B, Gibson CM, Pocock S, Huber K, Mehran R. Sex Differences Among Patients With High Risk Receiving Ticagrelor With or Without Aspirin After Percutaneous Coronary Intervention: A Subgroup Analysis of the TWILIGHT Randomized Clinical Trial. JAMA Cardiol. 2021 Sep 1;6(9):1032-1041. doi: 10.1001/jamacardio.2021.1720. PMID 33991416
- [Derived] Baber U, Dangas G, Angiolillo DJ, Cohen DJ, Sharma SK, Nicolas J, Briguori C, Cha JY, Collier T, Dudek D, Dzavik V, Escaned J, Gil R, Gurbel P, Hamm CW, Henry T, Huber K, Kastrati A, Kaul U, Kornowski R, Krucoff M, Kunadian V, Marx SO, Mehta S, Moliterno D, Ohman EM, Oldroyd K, Sardella G, Sartori S, Shlofmitz R, Steg PG, Weisz G, Witzenbichler B, Han YL, Pocock S, Gibson CM, Mehran R. Ticagrelor alone vs. ticagrelor plus aspirin following percutaneous coronary intervention in patients with non-ST-segment elevation acute coronary syndromes: TWILIGHT-ACS. Eur Heart J. 2020 Oct 1;41(37):3533-3545. doi: 10.1093/eurheartj/ehaa670. PMID 33085967
- [Derived] Dangas G, Baber U, Sharma S, Giustino G, Mehta S, Cohen DJ, Angiolillo DJ, Sartori S, Chandiramani R, Briguori C, Dudek D, Escaned J, Huber K, Collier T, Kornowski R, Kunadian V, Kaul U, Oldroyd K, Sardella G, Shlofmitz R, Witzenbichler B, Ya-Ling H, Pocock S, Gibson CM, Mehran R. Ticagrelor With or Without Aspirin After Complex PCI. J Am Coll Cardiol. 2020 May 19;75(19):2414-2424. doi: 10.1016/j.jacc.2020.03.011. Epub 2020 Mar 30. PMID 32240761
- [Derived] Angiolillo DJ, Baber U, Sartori S, Briguori C, Dangas G, Cohen DJ, Mehta SR, Gibson CM, Chandiramani R, Huber K, Kornowski R, Weisz G, Kunadian V, Oldroyd KG, Ya-Ling H, Kaul U, Witzenbichler B, Dudek D, Sardella G, Escaned J, Sharma S, Shlofmitz RA, Collier T, Pocock S, Mehran R. Ticagrelor With or Without Aspirin in High-Risk Patients With Diabetes Mellitus Undergoing Percutaneous Coronary Intervention. J Am Coll Cardiol. 2020 May 19;75(19):2403-2413. doi: 10.1016/j.jacc.2020.03.008. Epub 2020 Mar 30. PMID 32240760
- [Derived] Mehran R, Baber U, Sharma SK, Cohen DJ, Angiolillo DJ, Briguori C, Cha JY, Collier T, Dangas G, Dudek D, Dzavik V, Escaned J, Gil R, Gurbel P, Hamm CW, Henry T, Huber K, Kastrati A, Kaul U, Kornowski R, Krucoff M, Kunadian V, Marx SO, Mehta SR, Moliterno D, Ohman EM, Oldroyd K, Sardella G, Sartori S, Shlofmitz R, Steg PG, Weisz G, Witzenbichler B, Han YL, Pocock S, Gibson CM. Ticagrelor with or without Aspirin in High-Risk Patients after PCI. N Engl J Med. 2019 Nov 21;381(21):2032-2042. doi: 10.1056/NEJMoa1908419. Epub 2019 Sep 26. PMID 31556978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2015 through December 2017, 9006 patients were enrolled, and 7119 underwent randomization after 3 months
Pre-assignment Details: 1887 excluded from randomization (106 lost to follow up, 243 had adverse events between enrollment and randomization: a) myocardial infarction, stroke or death, b) revascularizations, and/or c) BARC type 3b or higher bleedings, 1148 were not adherent to DAPT, 267 withdrew consent or declined to participate, and 123 had other reasons.)
Period: Overall Study
Arm/Group | Placebo + Ticagrelor | Aspirin + Ticagrelor
Started | 3555 | 3564
Completed | 3496 | 3511
Not Completed | 59 | 53
Not completed — Withdrawal by Subject | 18 | 25
Not completed — Lost to Follow-up | 41 | 27
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Ticagrelor | Aspirin + Ticagrelor | Total
Number analyzed (Participants) | 3555 | 3564 | 7119
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (10.3) | 65.1 (10.4) | 65.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 846 | 852 | 1698
  Male | 2709 | 2712 | 5421
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Nonwhite race | 1110 | 1086 | 2196
  Unknown | 2445 | 2478 | 4923
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 1484 | 1488 | 2972
  Europe | 1251 | 1258 | 2509
  China | 512 | 516 | 1028
  India | 308 | 302 | 610
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (5.5) | 28.5 (5.6) | 28.6 (5.6)
Diabetes Mellitus [Count of Participants; unit: Participants] | 1319 | 1301 | 2620
Diabetes treated with Insulin [Count of Participants; unit: Participants] | 335 | 374 | 709
Chronic Kidney Disease (CKD) [Count of Participants; unit: Participants] — Population: multinational trial involving over 9000 patients across 187 sites - some variables were missing and not entered into the system in some of the sites. active efforts were made to retrieve these variables but in some cases it was not possible.
  Participants
    number analyzed (Participants) | 3410 | 3425 | 6835
    (all) | 572 | 573 | 1145
Anemia [Count of Participants; unit: Participants] — Population: multinational trial involving over 9000 patients across 187 sites - some variables were missing and not entered into the system in some of the sites. active efforts were made to retrieve these variables but in some cases it was not possible.
  Participants
    number analyzed (Participants) | 3405 | 3423 | 6828
    (all) | 675 | 654 | 1329
Current smoker [Count of Participants; unit: Participants] — Population: multinational trial involving over 9000 patients across 187 sites - some variables were missing and not entered into the system in some of the sites. active efforts were made to retrieve these variables but in some cases it was not possible.
  Participants
    number analyzed (Participants) | 3553 | 3562 | 7115
    (all) | 726 | 822 | 1548
Hypercholesterolemia [Count of Participants; unit: Participants] | 2157 | 2146 | 4303
Hypertension [Count of Participants; unit: Participants] — Population: multinational trial involving over 9000 patients across 187 sites - some variables were missing and not entered into the system in some of the sites. active efforts were made to retrieve these variables but in some cases it was not possible.
  Participants
    number analyzed (Participants) | 3554 | 3563 | 7117
    (all) | 2580 | 2574 | 5154
Peripheral Arterial Disease (PAD) [Count of Participants; unit: Participants] | 245 | 244 | 489
Previous Myocardial Infarction (MI) [Count of Participants; unit: Participants] | 1020 | 1020 | 2040
Previous Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants] | 1502 | 1496 | 2998
Previous Coronary Artery Bypass Graft (CABG) [Count of Participants; unit: Participants] — Population: multinational trial involving over 9000 patients across 187 sites - some variables were missing and not entered into the system in some of the sites. active efforts were made to retrieve these variables but in some cases it was not possible.
  Participants
    number analyzed (Participants) | 3554 | 3564 | 7118
    (all) | 362 | 348 | 710
Multivessel Coronary Artery Disease (CAD) [Count of Participants; unit: Participants] | 2272 | 2194 | 4466
Previous Major Bleeding Event [Count of Participants; unit: Participants] | 31 | 32 | 63
Indication for PCI [Count of Participants; unit: Participants] — Population: multinational trial involving over 9000 patients across 187 sites - some variables were missing and not entered into the system in some of the sites. active efforts were made to retrieve these variables but in some cases it was not possible.
  Participants
    Asymptomatic: number analyzed (Participants) | 3554 | 3563 | 7117
    Asymptomatic | 234 | 223 | 457
    Stable angina: number analyzed (Participants) | 3554 | 3563 | 7117
    Stable angina | 1047 | 999 | 2046
    Unstable angina: number analyzed (Participants) | 3554 | 3563 | 7117
    Unstable angina | 1249 | 1245 | 2494
    NSTEMI (non-ST-segment elevation MI): number analyzed (Participants) | 3554 | 3563 | 7117
    NSTEMI (non-ST-segment elevation MI) | 1024 | 1096 | 2120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With BARC Type 2, 3, or 5
Description: Number of participants with first occurrence of clinically relevant bleeding episode, defined as Bleeding Academic Research Consortium (BARC) Types 2, 3 or 5 bleeding. BARC bleeding types range from 0 (no bleeding) to 5 (fatal bleeding).
Time Frame: 12 months after randomization
Population: Data for the intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Ticagrelor | Aspirin + Ticagrelor
Number analyzed (Participants) | 3555 | 3564
Participants | 141 | 250

2. Secondary Outcome: Number of Participants With Ischemic Episode
Description: Number of participants with first occurrence of confirmed all-cause death, non-fatal myocardial infarction or stroke.
Time Frame: 12 months after randomization
Population: data for the per-protocol population , i.e., the participants who underwent randomization and had no major deviations from the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Ticagrelor | Aspirin + Ticagrelor
Number analyzed (Participants) | 3524 | 3515
Participants | 135 | 137

ADVERSE EVENTS:
Time Frame: 1 year
Description: All bleeding AE were reported in the intention-to-treat (ITT) cohort. - Placebo + Ticagrelor (N=3555) and Aspirin + Ticagrelor (N=3564)
  All ischemic AE were reported in the per protocol (PP) cohort. - Placebo + Ticagrelor (N=3524) and Aspirin + Ticagrelor (N=3515)
  All-cause mortality were reported in the per protocol (PP) cohort. - Placebo + Ticagrelor (N=3524) and Aspirin + Ticagrelor (N=3515)
Arm/Group | Placebo + Ticagrelor | Aspirin + Ticagrelor
All-Cause Mortality (participants affected / at risk) | 34/3524 | 45/3515
Serious Adverse Events (participants affected / at risk) | 262/3555 | 370/3564
Other Adverse Events (participants affected / at risk) | 0/3555 | 0/3564
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo + Ticagrelor (N=3555) | Aspirin + Ticagrelor (N=3564)
Myocardial Infarction (Cardiac disorders) | 95/3524 | 97/3515
Ischemic Stroke (Vascular disorders) | 18/3524 | 10/3515
Stent Thrombosis, definite or probable (Injury, poisoning and procedural complications) | 14/3524 | 20/3515
BARC 235 (Vascular disorders) | 141 | 250 — BARC type 2, 3, 5 bleeding

LIMITATIONS AND CAVEATS:
Limitations include lack of power to detect differences in the risk of important yet rare clinical events, e.g stent thrombosis and stroke; and trial may not be generalizable to all patients undergoing PCI due to high risk criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator remains responsible & has final approval for any publication and can publish/present results but shall submit manuscript/material proposed for publication/presentation relating to results to AZ for review ≤45 days prior to submission. AZ has 45 days to respond with comments. If requested by AZ, Investigator shall delay submission for further period ≤45 days, for deemed appropriate measures to establish/preserve parties' proprietary rights in intellectual property disclosed.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT02270242/Prot_SAP_001.pdf